CLINICAL TRIAL: NCT00370968
Title: Extended Studies on Safety and Efficacy of Zinc-ORS Compared to ORS Alone in Hospitalized Children With Severe and Complicated Acute Diarrhea
Brief Title: Zinc-ORS in Severe and Complicated Acute Diarrhea
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Centre For International Health (Other)
Collaborators: All India Institute of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IND-040 ICP (2001)/13
Record Dates: First submitted 2006-08-31; First posted 2006-09-01 (Estimated); Last update posted 2010-05-13 (Estimated); Status verified 2010-05

CONDITIONS: Diarrhea; Dehydration
Keywords: Children; India; Hospital; Zinc; Malnutrition; Treatment
MeSH Terms: conditions — Diarrhea; Dehydration; Malnutrition | interventions — Zinc Sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Zinc sulphate

SUMMARY:
Three-hundred-and-fifty-two males aged 1-36 months with acute non-dysenteric diarrhoea and no systemic illness will be enrolled in this clinical trial. Eligible children will be stratified by their age (1up to 5 months, 6-35 months). Within the two age strata the patients will be randomized to receive zinc-ORS (fortified with 40 mg elemental zinc as zinc gluconate per litre) or standard WHO ORS. The major outcome measures will be stool output and duration of diarrhea. The safety of administering zinc will be determined by examining the effect of zinc ingestion on vomiting, sodium and potassium homeostasis, plasma zinc and copper, and iron stores and concentration of serum transferrin receptor.

DETAILED DESCRIPTION:
Zinc deficiency is prevalent in developing countries due to inadequate food intake, low intake of foods from animal sources and high dietary intake of phytate, a substance that reduces zinc absorption. A recently completed trial at All India Institute Of Medical Sciences (AIIMS) measured the effect of zinc-ORS in the community, where most episodes are relatively mild. Zinc-ORS was efficacious in reducing the total number of stools (19% relative risk reduction, 95% CI 15% to 23%) and duration of diarrhoea (11% relative risk reduction, 95% CI 4% to 24%). In order to make policy decisions that standard ORS provided to children be fortified with zinc the national (and international) child health programs need a similar evidence base also for children hospitalized because of acute diarrhea. This is because these children represent the more severe end of the disease spectrum, i.e. they are the ones who are at the highest risk of dying.

The primary objective is to conduct a study of zinc-ORS in a hospital setting (i.e. of more severe diarrhea) to optimize and accurately measure the amount of zinc-ORS consumed and monitor stool output which is not possible in a field setting. The study will also examine the safety of using zinc-ORS; whether zinc-ORS affects the blood levels of sodium and potassium and of other micronutrients than zinc, such as copper and iron. The study will contribute to introducing a more efficacious ORS and help increase the ORS use rate which continues to be an important public health challenge in India.

The study will be carried out at two Clinical Research Facilities supervised by the Centre for Diarrhoeal Diseases and Nutrition Research, Division of Gastroenterology, Department of Pediatrics, AIIMS. 352 males aged 1-36 months with acute non-dysenteric diarrhoea and no systemic illness will be enrolled. Eligible children will be first stratified by their age (1up to 5 months, 6-35 months). Within the two age strata the patients will be randomized to receive zinc-ORS (fortified with 40 mg elemental zinc as zinc gluconate per litre) or standard WHO ORS. The major outcome measures will be stool output and duration of diarrhea. The safety of administering zinc will be determined by examining the effect of zinc ingestion on vomiting, sodium and potassium homeostasis, plasma zinc and copper, and iron stores and concentration of serum transferrin receptor. Minimum period of the study will be 48 hours and subjects will be discharged when diarrhoea has ceased or at 48 hours, whichever is later.

ELIGIBILITY:
Inclusion Criteria:

* Males
* Age 1 month up to 36 months:
* Passage of 3 or more liquid stools in a 24-hour period, every day, and at least one in 12 hours prior to admission
* Diarrhea for < 7days (168 hours)

Exclusion Criteria:

* severe systemic illness requiring intensive care management; systemic infection will be suspected if there is a general appearance of non-wellbeing with one or more of the following symptoms: shrill cry and irritability, temperature instability, hypotension, hypoglycemia, altered sensorium, lethargy or refusal of feeds, abdominal distension.
* chronic illness like Tuberculosis, Nephrotic syndrome, malignancy etc or any surgical disorder.
* severe malnutrition (weight for age <65% of NCHS median
* gross blood in stool
* refusal of consent

Ages: 1 Month to 36 Months | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 352
Dates: Start 2003-09; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Stool output (g/kg/24h)
Duration of diarrhoea (days).

CONTACTS AND LOCATIONS:
Overall Officials: Shinjini Bhatnagar, PhD, MBBS, Principal Investigator — All India Institute of Medical Sciences; Tor A Strand, MD, PhD, Study Chair — Centre For International Health; Halvor Sommerfelt, MD, PhD, Study Director — Centre For International Health
Locations (2):
- India (2):
  - All India Institute of Medical Sciences, New Delhi
  - Deen Dayal Upadhyaya Hospital, New Delhi

REFERENCES:
- [Background] Strand TA, Chandyo RK, Bahl R, Sharma PR, Adhikari RK, Bhandari N, Ulvik RJ, Molbak K, Bhan MK, Sommerfelt H. Effectiveness and efficacy of zinc for the treatment of acute diarrhea in young children. Pediatrics. 2002 May;109(5):898-903. doi: 10.1542/peds.109.5.898. PMID 11986453
- [Background] Mahalanabis D, Chowdhury A, Jana S, Bhattacharya MK, Chakrabarti MK, Wahed MA, Khaled MA. Zinc supplementation as adjunct therapy in children with measles accompanied by pneumonia: a double-blind, randomized controlled trial. Am J Clin Nutr. 2002 Sep;76(3):604-7. doi: 10.1093/ajcn/76.3.604. PMID 12198006
- [Background] Mahalanabis D, Bhan MK. Micronutrients as adjunct therapy of acute illness in children: impact on the episode outcome and policy implications of current findings. Br J Nutr. 2001 May;85 Suppl 2:S151-8. doi: 10.1079/bjn2000308. PMID 11509104
- [Background] Fontaine O. Effect of zinc supplementation on clinical course of acute diarrhoea. J Health Popul Nutr. 2001 Dec;19(4):339-46. PMID 11855358
- [Background] Brooks WA, Santosham M, Roy SK, Faruque AS, Wahed MA, Nahar K, Khan AI, Khan AF, Fuchs GJ, Black RE. Efficacy of zinc in young infants with acute watery diarrhea. Am J Clin Nutr. 2005 Sep;82(3):605-10. doi: 10.1093/ajcn.82.3.605. PMID 16155274
- [Background] Bahl R, Bhandari N, Saksena M, Strand T, Kumar GT, Bhan MK, Sommerfelt H. Efficacy of zinc-fortified oral rehydration solution in 6- to 35-month-old children with acute diarrhea. J Pediatr. 2002 Nov;141(5):677-82. doi: 10.1067/mpd.2002.128543. PMID 12410197
- [Background] Baqui AH, Black RE, El Arifeen S, Yunus M, Chakraborty J, Ahmed S, Vaughan JP. Effect of zinc supplementation started during diarrhoea on morbidity and mortality in Bangladeshi children: community randomised trial. BMJ. 2002 Nov 9;325(7372):1059. doi: 10.1136/bmj.325.7372.1059. PMID 12424162
- [Background] Bhandari N, Bahl R, Taneja S, Strand T, Molbak K, Ulvik RJ, Sommerfelt H, Bhan MK. Substantial reduction in severe diarrheal morbidity by daily zinc supplementation in young north Indian children. Pediatrics. 2002 Jun;109(6):e86. doi: 10.1542/peds.109.6.e86. PMID 12042580
- [Background] Sazawal S, Black RE, Bhan MK, Bhandari N, Sinha A, Jalla S. Zinc supplementation in young children with acute diarrhea in India. N Engl J Med. 1995 Sep 28;333(13):839-44. doi: 10.1056/NEJM199509283331304. PMID 7651474
- [Derived] Wadhwa N, Natchu UC, Sommerfelt H, Strand TA, Kapoor V, Saini S, Kainth US, Bhatnagar S. ORS containing zinc does not reduce duration or stool volume of acute diarrhea in hospitalized children. J Pediatr Gastroenterol Nutr. 2011 Aug;53(2):161-7. doi: 10.1097/MPG.0b013e318213ca55. PMID 21788757